CLINICAL TRIAL: NCT06756256
Title: The Effect of Wearing Customized Insole on Foot Alignment, Body Alignment, and Balance Ability in Stroke Patients
Brief Title: Effect of Foot Insole on Body Alignment, and in Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Meeyoung Kim, Assistant Professor, University of Sharjah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WonkwangUoS
Record Dates: First submitted 2024-12-25; First posted 2025-01-01 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Stroke
Keywords: Stroke; Insole; Foot arch; Body alignment; Balance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: A prospective, double-blinded, parallel, randomized clinical trial. 20 participants will be divided into 2 groups, intervention and control group. 10 will be in the intervention group that will wear the customized insole for 6 weeks whereas the 10 others will not during the same period of time.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants and outcome assessors will be blinded to the treatment methods and group allocation. Assessor blinding will be obtained through an independent research assist: not knowing the study design and not specifically involved in any other aspect of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3D Insole (Experimental): Intervention group who will wear the customized insole for 6 weeks during daily activities. Insole production will be through the following process.
  The participants' feet will be visually inspected for abnormalities, and the MediAce Scanner-MS320F will scan the feet in a seated position with the knees and ankles fixed at 90°. MediAce Scanner-MS320F's software will automatically calculate and correct the anatomical position of bones and joints. The corrected models will produce the printed insoles.
  Apart from wearing insole, they will receive the physiotherapy treatment as their continuation of rehabilitation program.
  Interventions: Device: Customized insole
- Control_without 3D Insole (No Intervention): Participants in the control group will not wear the customized insoles for 6 weeks. They will receive the physiotherapy treatment as their continuation of rehabilitation program.

INTERVENTIONS:
Device: Customized insole — Participants will wear the produced customized insoles during daily activities and interventions for six weeks under the guidance of physical therapists working at Miso Hospital in Iksan City. As their continuation of their rehabilitation program, they will receive a conservative physiotherapy treatment five times a week for six weeks.
  Other Names: Insole made by MediAce Scanner-MS320F
  Arms: 3D Insole

SUMMARY:
Goal: This study will be conducted to find out the effects of customized insole on foot alignment, body alignment, and balance ability of stroke patients.

Recruitment: Total 20 participants will be recruited and will be divided into 2 groups: Intervention and control group with or without wearing foot insole for 6 weeks.

Evaluation tool:

1. MediACE Scanner-MS320F will be used to evaluate foot alignment and will create customized insole.
2. Exbody 770 will be used to measure body alignment.
3. Timed up & go test will be used to evaluate dynamic balance.

Intervention: The intervention group will wear a customized insole during daily life for 6 weeks whereas the control group will not.

Evaluation will be conducted 2 times before and after 6 weeks.

DETAILED DESCRIPTION:
This study will recruit 20 stroke patients and will randomly assign them to the intervention group (n=10) and control group (n=10). After given the full description of the study, participants who will voluntarily agreed to participate will be included.

This study involves producing customized insoles for participants to wear during daily activities for six weeks. The customized insoles will be produced using the MediAce Scanner-MS320F, which scans the participants' feet in a seated position.

The participants in the intervention group will wear the produced insoles during daily activities. Their rehabilitation program will be continued apart from the insole wearing.

The participants in the control group will wear their normal insoles during daily activities. Also, their rehabilitation program will be continues as same as the intervention group.

Outcome measure will be conducted twice, pre- and post-intervention. It includes foot alignments and arch height using the MediACE Scanner-MS320F, body alignments using the Exbody 770, and balance ability using the Timed Up & Go test.

ELIGIBILITY:
Inclusion Criteria:

* Chronic (more than 1 year ago) stroke patient over 50 years old
* MMSE (mini-mental state examination) score of 24 or higher out of 30, capable of understanding the experimenter's instructions
* No history of orthopedic surgery
* Voluntarily agreed to participate

Exclusion Criteria:

* Neurological problems other than stroke affecting balance ability
* Movement restrictions or involuntary limb movements due to ankle pain
* Severe visual impairment, field defects, cognitive impairment making it impossible to use evaluation equipment
* Taking medication affecting posture and balance ability

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
Foot alignment | Outcome measure will be done twice before and after 6 weeks' intervention period.
  Foot alignment will be measured with 3 parameters including medial longitudinal arch angle, transverse arch angle, and arch height. Measurement will be performed by MediACE Scanner-MS320F (Real Dimension Co., South Korea).
  Outcome measure will be done twice before and after 6 weeks' intervention period as below. The MediACE Scanner-MS320F analyzes anatomical information of the leg by applying a marker recognition algorithm to 15 bones and joints of the foot, measuring angles and heights of the medial longitudinal arch, transverse arch, medial malleolus, and navicular bone tuberosity.
Body alignment | Outcome measure will be done twice before and after 6 weeks' intervention period.
  Body alignment will be measured with 3 parameters including shoulder tilt angle, pelvic tilt angle, and knee tilt angle. Measurement will be conducted by Exbody 770 (Exbody Co., South Korea) before and after 6 weeks' intervention period as following procedure.
  The Exbody 770 identifies joints automatically with an infrared camera, examines musculoskeletal misalignment and imbalance, and visually confirms body alignment by displaying the condition of the cervical, lumbar, knee, and ankle joints in 3D from the front and side.
Timed Up & Go | Outcome measure will be done twice before and after 6 weeks' intervention period.
  The Timed Up & Go test will be used to measure balance ability before and after 6 weeks' intervention period. Procedure description is as below.
  Participants, wearing comfortable shoes, rise from a chair with armrests, walk 3 meters, turn around, and sit back down, timed without assistance. The average of three trials will be used as their balance ability.

CONTACTS AND LOCATIONS:
Overall Officials: Meeyoung Kim, Principal Investigator — University of Sharjah
Locations (1):
- Wonkwang Health Science University, Iksan, Jeolla, South Korea

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol, SAP
Time Frame: After 6 months of completing a study and available for one year
Access Criteria: Not identified yet

REFERENCES:
- [Background] Wang J, Qiao L, Yu L, Wang Y, Taiar R, Zhang Y, Fu W. Effect of Customized Insoles on Gait in Post-Stroke Hemiparetic Individuals: A Randomized Controlled Trial. Biology (Basel). 2021 Nov 15;10(11):1187. doi: 10.3390/biology10111187. PMID 34827179
- [Background] Hozein M, Mortada H, Hamed M, Abdelhaleem N, Elshennawy S. Effect of insole on postural control and gait of stroke patients: a systematic review and meta-analysis. Int J Rehabil Res. 2024 Sep 1;47(3):137-146. doi: 10.1097/MRR.0000000000000632. Epub 2024 Jun 17. PMID 38881488
- [Background] Liu YT, Tsai HT, Hsu CY, Lin YN. Effects of orthopedic insoles on postural balance in patients with chronic stroke: A randomized crossover study. Gait Posture. 2021 Jun;87:75-80. doi: 10.1016/j.gaitpost.2021.04.014. Epub 2021 Apr 20. PMID 33894465
- [Background] Ma CC, Rao N, Muthukrishnan S, Aruin AS. A textured insole improves gait symmetry in individuals with stroke. Disabil Rehabil. 2018 Nov;40(23):2798-2802. doi: 10.1080/09638288.2017.1362477. Epub 2017 Aug 7. PMID 28783984
- [Background] Fu JC, Chen YJ, Li CF, Hsiao YH, Chen CH. The effect of three dimensional printing hinged ankle foot orthosis for equinovarus control in stroke patients. Clin Biomech (Bristol). 2022 Apr;94:105622. doi: 10.1016/j.clinbiomech.2022.105622. Epub 2022 Mar 11. PMID 35325715